CLINICAL TRIAL: NCT02350478
Title: Effects of Linagliptin on Endothelial Function and Global Arginine Bioavailability Ratio in Coronary Artery Disease Patients With Early Diabetes
Brief Title: Effects of Linagliptin on Endothelial Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-2012-01
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Type 2 Diabetes; Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — Linagliptin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Linagliptin (Active Comparator): The subjects will receive Linagliptin 5mg (licensed dose for treatment of type 2 diabetes) .
  Interventions: Drug: Linagliptin
- Placebo (Placebo Comparator): The subjects will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linagliptin — The subject will receive Linagliptin 5mg orally once daily for 12 weeks.
  Other Names: Trajenta
  Arms: Linagliptin
Drug: Placebo — The subject will receive placebo orally once daily for 12 weeks.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
This study is planned to evaluate if linagliptin can improve endothelial function in patients with type 2 diabetes mellitus. In addition, the effect of linagliptin on arginine bioavailability ratios and postchallenge glycaemic control will be studied.

DETAILED DESCRIPTION:
Patients with type 2 diabetes (T2DM) are at increased risk of macrovascular events as well as microvascular complications. It is well known, that the pathophysiologic process of type 2 diabetes starts many years before the diagnosis can be made on the basis of elevated fasting blood glucose. In particular the data of the United Kingdom Prospective Diabetes Study (UKPDS) study and the UKPDS post trial monitoring highlighted the importance of an early glucose lowering intervention in patients with T2DM with respect to micro- and macrovascular complications. The investigators and in particular the Euro Heart survey on Diabetes and the Heart demonstrated, that in a cardiovascular high risk population, namely patients with coronary artery disease (CAD), about 35% suffer from manifest type 2 diabetes. In addition, another 9 to 15% of CAD patients have postchallenge diabetes, diagnosed on the basis of an oral glucose tolerance test, which means that approximately a half of all patients with CAD have diabetes.

Recently the investigators could demonstrate that not only established type 2 diabetes diagnosed on the basis of fasting hyperglycaemia is associated with an increased cardiovascular risk, but also postchallenge hyperglycemia (i.e. impaired glucose tolerance or postchallenge diabetes).

Dipeptidylpeptidase-4 (DPP-4) inhibitors increase endogenous glucagon like-peptide-1 (GLP-1) levels and GLP-1 in turn increases the insulin release from pancreatic beta-cells in a glucose dependent manner as well as suppresses glucagon secretion from pancreatic alpha cells. Investigations in type 2 diabetic patients showed that this drug class lowers both, fasting and postchallenge or postmeal glucose levels and hence, HbA1c and is well tolerated.

However, the lowering of the surrogate measurement HbA1c has not necessarily turned out to translate into a reduced number of cardiovascular events in patients with T2DM. In contrary in particular for the thiazolidinedione Rosiglitazone concerns about an increased risk of cardiovascular events have been raised despite a robust HbA1c lowering effect.Therefore the Food and Drug Administration (FDA) and the European Medicines Agency (EMA) issued in 2008 and 2010, respectively, guidance for new glucose lowering drugs, requiring proof of at least cardiovascular safety. Cardiovascular outcome trials with Linagliptin are currently being performed (CAROLINA, CARMELINA), however, it will take a couple of years until the results are available.A well known and validated cardiovascular surrogate parameter is endothelial dysfunction. The investigators and others have shown previously, that endothelial dysfunction is present in patients with coronary artery disease and early diabetes and can be improved by pharmacological intervention. This surrogate measurement could be helpful in better understanding the cardiovascular effects of Linagliptin while awaiting the results of the definitive outcome trials.

The aim of this study is to investigate the effects of Linagliptin in coronary patients with early T2DM on various cardiovascular surrogate measurements including mechanical and biochemical endothelial function assessments. The overarching aim of our study is to investigate the effects of Linagliptin on endothelial function, arginine bioavailability ratios and postchallenge glycaemic control in patients with early diabetes and coronary atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 to 80 years
* Early diabetes (postchallenge diabetes (2h glucose >200 mg/dl or type 2 diabetes treated with diet only or on a stable dose of metformin monotherapy)
* Coronary atherosclerosis (diagnosed via coronary angiography or coronary computer tomography)

Exclusion Criteria:

* Acute coronary syndrome or cerebrovascular event within the previous 4 weeks
* Body Mass Index (BMI) > 35 kg/m2
* HbA1c <6.0% (42 mmol/mol)
* Serum creatinine > 2.5 mg/dl
* Aspartate Transaminase (AST)/Alanine Transaminase (ALT)>3x upper limit of normal
* HbA1c >9.0% (>75 mmol/mol)
* Heart failure > New York Heart Association (NYHA) class II
* Uncontrolled hypertension (blood pressure > 165 / 100 mmHg)
* Treatment with orally administered steroids
* New onset statin or Angiotensin Converting Enzym- (ACE-) inhibitor within the previous 6 weeks
* Known Malignancy
* Pregnancy or breast feeding women.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-07; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harald Sourij, Assoc.-Prof., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Department for Internal Medicine, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tripolt NJ, Aberer F, Riedl R, Url J, Dimsity G, Meinitzer A, Stojakovic T, Aziz F, Hodl R, Brachtl G, Strunk D, Brodmann M, Hafner F, Sourij H. Effects of linagliptin on endothelial function and postprandial lipids in coronary artery disease patients with early diabetes: a randomized, placebo-controlled, double-blind trial. Cardiovasc Diabetol. 2018 May 17;17(1):71. doi: 10.1186/s12933-018-0716-x. PMID 29773079
- [Derived] Tripolt NJ, Aberer F, Riedl R, Hutz B, Url J, Dimsity G, Meinitzer A, Stojakovic T, Hodl R, Brodmann M, Hafner F, Sourij H. The effects of linagliptin on endothelial function and global arginine bioavailability ratio in coronary artery disease patients with early diabetes: study protocol for a randomized controlled trial. Trials. 2016 Oct 13;17(1):495. doi: 10.1186/s13063-016-1627-3. PMID 27733180

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Linagliptin | Placebo
Started | 25 | 24
Completed | 20 | 23
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Linagliptin | Placebo | Total
Number analyzed (Participants) | 20 | 23 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (7.8) | 63.3 (8.7) | 63.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 15 | 19 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 23 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 20 | 23 | 43
Blood pressure systolic (mmHg) [Mean (Standard Deviation); unit: mmHg] | 134 (17) | 128 (18) | 131 (18)
Blood pressure diastolic (mmHg) [Mean (Standard Deviation); unit: mmHg] | 79 (14) | 78 (10) | 79 (12)
Low density lipoprotein (mg/dl) [Mean (Standard Deviation); unit: mg/dl] | 66 (31) | 76 (43) | 71 (37)
Triglycerides (mg/dl) [Median (Inter-Quartile Range); unit: mg/dl] | 145 [54 to 480] | 122 [63 to 255] | 128 [90 to 163]
HbA1c (mmol/mol) [Median (Inter-Quartile Range); unit: mmol/mol] | 50.5 [43 to 69] | 51 [39 to 78] | 51 [45.5 to 55.5]
Fasting blood glucose [Mean (Standard Deviation); unit: mg/dl] | 136 (41) | 123 (26) | 135 (35)
Aspartate-Aminotransferase (U/L) [Mean (Standard Deviation); unit: U/l] | 33.5 (14) | 27.6 (8.3) | 30.4 (11.6)
Alanine-Aminotransferase (U/L) [Mean (Standard Deviation); unit: U/l] | 40.4 (25) | 29 (12.7) | 34.4 (20.1)
Creatinine (mg/dL) [Mean (Standard Deviation); unit: mg/dl] | 1.0 (0.3) | 1.0 (0.2) | 1.0 (0.3)
estimated glomerular filtration rate (ml/min) [Mean (Standard Deviation); unit: ml/min] | 76.7 (16.1) | 80.8 (18.0) | 78.9 (17.0)
c-reactive protein (mg/L) [Mean (Standard Deviation); unit: mg/dl] | 3.8 (4.2) | 7.6 (20.4) | 5.8 (15.2)
Urine albumine´(mg/L) [Mean (Standard Deviation); unit: mg/l] | 51.8 (68.1) | 30.3 (43.4) | 40.8 (57.1)
n-terminal-proBNP (pg/ml) [Mean (Standard Deviation); unit: pg/ml] | 419 (528) | 228 (452) | 317 (492)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Endothelial Function (FMD - Flow Mediated Dilatation) From Baseline to 12 Weeks
Description: Endothelium-dependent FMD following reactive hyperaemia was examined in the brachial artery according to the guidelines described by Coretti et al (J Am Coll Cardiol. 2002;39(2):257-65). FMD-diameter is calculated as the average of the three diameter measurements following reactive hyperaemia. FMD was calculated as the percent change in diameter compared to baseline. Flow-mediated dilation is reported such as "percentage of change in diameter (%)".
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of change in diameter (%)
Arm/Group | Linagliptin | Placebo
Number analyzed (Participants) | 20 | 23
percentage of change in diameter (%) | 0.4 (4.8) | -0.5 (3.0)

2. Secondary Outcome: Changes in Global Arginine Bioavailability Ratio (Ratio of Arginine to [Ornithine + Citrulline]) and Arginine to Ornithine Ratio From Baseline to 12 Weeks
Description: Arginine, ornithine and citrulline will be measured in serum samples with a conventional usual amino acid analysis technique, involving separation of amino acids by ion exchange chromatography followed by postcolumn continuous reaction with ninhydrin. Global arginine bioavailability ratio (GABR) will be calculated by L-arginine divided by the sum of (L-ornithine plus L-citrulline). The arginine to ornithine ratio will be calculated by dividing L-arginine by L-ornithine levels.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Linagliptin | Placebo
Number analyzed (Participants) | 20 | 23
Ratio
  Global Arginine Bioavailabilty Ratio (%) | -0.11 (0.35) | -0.06 (0.39)
  Arginine to ornithine ratio (%) | -0.13 (0.45) | -0.05 (0.53)

3. Secondary Outcome: Changes in Biochemical Markers (sICAM-1)
Description: Soluble cell adhesion molecules-1 (sICAM-1) of endothelial function from baseline to 12 weeks
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Linagliptin | Placebo
Number analyzed (Participants) | 20 | 23
ng/ml | -15 [-272 to 103] | -21 [-134 to 310]

4. Secondary Outcome: Changes in the Area Under Curve (AUC) of Glucose, Insulin and C-peptide During the Meal Tolerance Test From Baseline to 12 Weeks
Description: The Area under the curve was calculated for glucose, insulin and for the free fatty acids based on the trapezoidal rule with baseline value as the mean of the values at time points -5 and 0 minutes.
  The Meal Tolerance Test (MTT) was performed after an overnight fast (apart from water). A pre-meal blood sample will be taken (-5mins) and then all subjects will be asked to drink Fortimel compact (10 kcal/kg) over a period of 2-4 mins (time 0 mins). During the mixed meal test further blood samples will be taken at 15, 30, 60, and 120 minutes. All samples will be used for the determination of glucose, insulin and free fatty acids. The blood at each time point will be placed into a fluoride oxalate tube (1ml) for plasma glucose and into a serum tube for insulin and free fatty acids.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg*min/dl
Arm/Group | Linagliptin | Placebo
Number analyzed (Participants) | 20 | 23
mg*min/dl
  Glucose AUC | -1135 (2619) | 481 (3185)
  C-peptide AUC | -3 (161) | -34 (211)
  Insulin AUC | 249 (4766) | 40 (6357)

5. Secondary Outcome: Changes in the Area Under Curve (AUC) of Free Fatty Acids During the Meal Tolerance Test From Baseline to 12 Weeks
Description: The Area under the curve was calculated for glucose, insulin and for the free fatty acids based on the trapezoidal rule with baseline value as the mean of the values at time points -5 and 0 minutes.
  The MTT was performed after an overnight fast (apart from water). A pre-meal blood sample will be taken (-5mins) and then all subjects will be asked to drink Fortimel compact (10 kcal/kg) over a period of 2-4 mins (time 0 mins). During the mixed meal test further blood samples will be taken at 15, 30, 60, and 120 minutes. All samples will be used for the determination of glucose, insulin and free fatty acids. The blood at each time point will be placed into a fluoride oxalate tube (1ml) for plasma glucose and into a serum tube for insulin and free fatty acids.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: µmol*min/l
Arm/Group | Linagliptin | Placebo
Number analyzed (Participants) | 20 | 23
µmol*min/l | 2.0 (28.4) | -3.1 (18.3)

6. Secondary Outcome: Changes in Biochemical Markers (svCAM-1)
Description: Soluble cell adhesion molecules-1 (svCAM-1) of endothelial function from baseline to 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Linagliptin | Placebo
Number analyzed (Participants) | 20 | 23
ng/ml | -34 (84) | 5 (130)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 16 weeks (12 weeks of intervention and 4 weeks of follow-up).
Arm/Group | Linagliptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 3/20 | 1/23
Other Adverse Events (participants affected / at risk) | 2/20 | 3/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linagliptin (N=20) | Placebo (N=23)
discus prolaps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Borreliosis (Infections and infestations) | 0 (0) | 1 (1)
Coordinating disorders (Nervous system disorders) | 1 (1) | 0 (0) — Hospitalization due to coordinating disorders
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Hospitalisation due to abdominal pain
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linagliptin (N=20) | Placebo (N=23)
Dorsal pain (Nervous system disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Claudicatio intermittens (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2014-10-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT02350478/Prot_000.pdf